CLINICAL TRIAL: NCT05594264
Title: Developing and Implementing a Storytelling Intervention for African Americans Living With Hypertension
Brief Title: Storytelling Intervention for African Americans Living With Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended before the second phase of the study could be started. Additionally, the second phase of the study will be a part of the PIs K01 study.
Sponsor: University of Delaware (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1766419-7; 2P20GM113125-06 (NIH)
Record Dates: First submitted 2022-08-31; First posted 2022-10-26 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-06

CONDITIONS: Hypertension
Keywords: Storytelling; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The two phase study, included a feasibility phase. During the feasibility phase 30 participants would be recruited to provide feedback on the design of the website, the impact of the study, and preferences for future study designs. The second phase of the study was the pilot study. The objective of the 6-week study was to explore the impact of a web-based storytelling program on medication adherence and blood pressure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot Study (Experimental): The objective of the second phase of the study was to conduct a 6-week pilot study of the web-based storytelling approach
  Interventions: Behavioral: HBPStories
- Feasibility Phase (No Intervention): The objective of the feasibility phase was to assess participant views of the stories and the study website, and obtain feedback for the design of a future trial.

INTERVENTIONS:
Behavioral: HBPStories — The objective of this arm was to pilot test the web-based storytelling program to determine the preliminary impact on blood pressure and medication adherence, and if the web-based approach was an engaging approach for individuals managing hypertension.
  Arms: Pilot Study

SUMMARY:
Narrative communication (e.g., storytelling) is an approach that has contributed to behavioral change for individuals with conditions such as diabetes, breast cancer, and hypertension. The objective of this study is to conduct a feasibility and pilot study storytelling intervention for African Americans with hypertension. In the feasibility phase 30 African Americans with hypertension will be recruited to view nine patient stories and provide feedback on the effectiveness, usefulness, and satisfaction with the stories. Nine African Americans adults with hypertension were filmed, sharing experiences living with and managing hypertension; including, diet and exercise tips, suggestions for locating healthy foods, and motivational stories about successfully controlling hypertension. During the feasibility phase feedback will also be elicited from the participants about the best approaches for delivering a storytelling intervention, and obtain feedback on the resources and health information that would be helpful to an individual participating in a storytelling intervention. In the pilot study phase, 30 African Americans adults with hypertension will be recruited to participate in a 6-week trial, each week the participants will watch one story and review one module of health information accessible through the study specific website developed for the High Blood Pressure Stories (HBPStories) study. Data will be collected at baseline and 6-weeks including systolic and diastolic blood pressure, medication adherence, health behaviors such as diet and physical activity, and psychosocial measures including positive affect and self-efficacy in the management of hypertension.

ELIGIBILITY:
Inclusion Criteria:

The study inclusion criteria are as follows:

* self-reported hypertension
* race/ethnicity: Black or African American
* prescribed antihypertensive medication
* age ≥ 18 years

Exclusion Criteria:

The exclusion criteria are:

* cognitive limitations that limit the ability to provide informed consent
* unable to speak or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be available one year after the last participant is recruited. Study protocol, informed consent, and study surveys will be available immediately after recruitment is completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified study data will become available one year after the last participant is recruited, and will be available for three years. Supporting information will be available as soon as recruitment is completed.
Access Criteria: Please email the PI for access to study data and supporting information.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not recruited for the pilot study phase of the study.
Groups:
- Pilot Study Phase: 6-week trial of the web-based storytelling study
- Feasibility Phase: The objective of the feasibility phase of the study was to recruit 30 participants to view the video stories and provide feedback on engagement and satisfaction with the stories and recommendations for the design of a future research study.
Period: Overall Study
Arm/Group | Pilot Study Phase | Feasibility Phase
Started | 0 | 31
Completed (Pilot phase was not initiated, participants were not recruited for this phase of the study.) | 0 | 0
Not Completed | 0 | 31

BASELINE CHARACTERISTICS:
Population: Due to the delay in recruiting for the feasibility phase of the study, we were unable to conduct the 6-week trial. The PI was funded for a K01 and has incorporated the 6-week trial into the design of the K01 research.
Groups:
- Pilot Study: Participants will participate in a 6-week web-based storytelling study. A 6-week web-based study. Systolic blood pressure, diastolic blood pressure, and medication adherence will be measured at baseline and 6-weeks.
- Feasibility Study: Participants were invited to provide feedback on the effectiveness of the storytellers, engagement with the website and health information, and preferences for the design of a future intervention.
- Total: Total of all reporting groups
Arm/Group | Pilot Study | Feasibility Study | Total
Number analyzed (Participants) | 0 | 31 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 25 | 25
  >=65 years | 0 | 6 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 53 (15) | 53 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 26 | 26
  Male |  | 5 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education [Count of Participants; unit: Participants]
  some HS, HS, GED |  | 2 | 2
  Some College, Trade, Associates |  | 12 | 12
  Bachelors |  | 9 | 9
  Masters/Doctorate |  | 8 | 8
Income [Count of Participants; unit: Participants]
  <$50,000 |  | 18 | 18
  $50,000-<$100,000 |  | 8 | 8
  >$100,000 |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Description: Systolic and Diastolic Blood Pressure, Unit of Measure: Percentage of Individuals with Elevated or High Blood Pressure
Time Frame: 6 weeks
Population: Blood pressure was an outcome measure for the pilot study only. The pilot study was not initiated due to the funding ending before the study could begin. Blood pressure was not collected for either arm and there was no data to assess.
Groups:
- Feasibility Arm: The objective of the feasibility phase was to recruit 30 adults with hypertension to provide feedback on their engagement with the stories and the storyteller, the design of the study website, and share their preferences for future storytelling interventions.
Arm/Group | Pilot Study | Feasibility Arm
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Medication Adherence
Description: Self-reported medication adherence, Unit of Measure: Percentage of Individuals reporting low, moderate, or high adherence
Time Frame: 6 weeks
Population: Medication adherence was an outcome for the pilot study, not the feasibility study. The pilot study was not initiated due to the end of funding. Medication adherence data was not collected for any participants and there was no data to analyze.
Arm/Group | Pilot Study | Feasibility Arm
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Effectiveness and Engagement
Description: Effectiveness and engagement were measured in the cross-section survey for the feasibility phase of the study. These measures were used to explore participants perceptions of the stories, participants self reported if the stories were engaging and effective in promoting lifestyle change.
Time Frame: baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: There were two phases of the study, the feasibility phase and the pilot study. During the feasibility phase participants viewed the website and stories, and completed surveys during one visit. Adverse events were collected within 24 hours of participating in the feasibility phase. The second phase, the pilot study was not initiated due to funding ending; therefore, no adverse events were collected.
Description: The definition of adverse events or serious adverse events does not differ from the clinicaltrials.gov definition.
Groups:
- Pilot Study: Participants will participate in a 6-week web-based storytelling study. Systolic blood pressure, diastolic blood pressure, and medication adherence will be measured at baseline and 6-weeks.
- Feasibility Phase: Participants will review study website and stories, and provide feedback on effectiveness of the stories, engagement with the website, and preferences for lifestyle intervention study design.
Arm/Group | Pilot Study | Feasibility Phase
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/31
Other Adverse Events (participants affected / at risk) | 0/0 | 0/31

LIMITATIONS AND CAVEATS:
Recruitment for the feasibility study was delayed and we were able to recruit participants for the first phase of the study. The second phase of the study was not completed, the 6-week trial. However, the study was recently funded and the 6 week trial will be conducted as a part of a pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT05594264/Prot_000.pdf